CLINICAL TRIAL: NCT00793351
Title: Allogeneic Hematopoietic Stem Cell Transplantation With Reduced-intensity Conditioning in Children With Neuroblastoma Who Have Failed a Prior Autologous Transplantation
Brief Title: Reduced Intensity Stem Cell Transplantation in Children With Relapsed Neuroblastoma After Autologous Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Ki Woong Sung, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-08-073
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2015-11

CONDITIONS: Neuroblastoma
Keywords: reduced intensity stem cell transplantation for neuroblastoma; relapsed neuroblastoma after high-dose chemotherapy and autologous stem cell rescue
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Reduced-intensity allogeneic hematopoietic stem cell transplantation — Treatment Scheme
  * Enrollment - Pre-RIST treatment - RIST
  * 4 cycles of conventional chemotherapy will be given prior to RIST.
  * Surgery will be done whenever possible prior to RIST.
  * Local radiotherapy will be applied whenever possible prior to RIST.
  * topotecan + cyclophosphamide) regimen will be used for pre-RIST conventional chemotherapy.
  * Cyclophosphamide/Fludarabine (CyFlu) regimen will be used as conditioning regimen for matched related or unrelated SCT. CyFlu-ATG regimen will be used as conditioning regimen for mismatched related SCT.

SUMMARY:
The purpose of this study is to evaluate the feasibility and efficacy of reduced-intensity allogeneic stem cell transplantation (RIST) with RIC regimen in children with neuroblastoma who have failed a prior autologous stem cell transplantation. The investigators will investigate the potential of RIC regimen in inducing antitumor response if the present protocol will indeed reduce the early TRM and allow for sustained donor chimerism.

DETAILED DESCRIPTION:
The prognosis of high-risk neuroblastoma (NB) after conventional chemoradiotherapy is very poor. Therefore, a strategy using high-dose chemotherapy and autologous stem cell transplantation (HDCT/auto-SCT) has been explored to improve the prognosis of patients with high-risk NB. The results of randomized trials comparing HDCT/auto-SCT with chemotherapy alone showed a better event-free survival (EFS) in the auto-SCT arm than in the continuous chemotherapy arm. However, the overall EFS was still unsatisfactory. In this context, investigators have examined the efficacy of double or triple tandem auto-SCT to further improve the outcome of high-risk NB patients. George et al. carried out a single arm trial of tandem auto-SCT as consolidation therapy, and reported improved long-term survival (5-year progression-free survival 47%) with acceptable toxicity. Kletzel et al. also conducted a single arm trial of triple tandem auto-SCT and reported improved survival (3-year EFS 57%). Investigators in the present study also carried out tandem auto-SCT as consolidation therapy, and reported improved long-term survival (5-year progression-free survival 62%) with acceptable toxicity. However, unfortunately, tumor relapses in many patients even after tandem auto-SCT.

The major cause of treatment failure following auto-SCT remains relapse of the underlying disease. Additional chemotherapy after relapse in these patients have been ineffective, and therefore, new treatment strategies are warranted. In this context, allogeneic stem cell transplantation (allo-SCT) has been tried as salvage treatment in patients with NB who have failed a prior auto-SCT. Allo-SCT would theoretically be preferable in term of relapse-free survival because this has an antitumor effect due to a graft versus tumor (GVT) effect which is absent in auto-SCT. The graft versus leukemia (GVL) effect represents a widely accepted major component of allo-SCT, and there is emerging evidence also for a GVT effect in solid tumor. GVT effect was also demonstrated in patient with advanced NB who received HLA haplo-identical allo-SCT.

Generally, allo-SCT carries a lower risk of relapse, However, it has a much higher early treatment-related mortality (TRM) compared to auto-SCT. TRM rate in allo-SCT is especially high in patients who have failed a prior auto-SCT. The 1-year TRM rate following a conventional (ie myeloablative) allo-SCT in adult recipients of a prior auto-SCT has been reported as high as 50-85%. In children, transplantation-related toxicity was also one of the major obstacles in conventional allo-SCT because they had been already heavily treated prior to allo-SCT. Therefore, this salvage strategy has showed a limited success in the majority of children with relapsed NB who have failed a prior single or tandem auto-SCT, although allo-SCT is supposed to be the only curative treatment in patients. Only a small proportion of these patients have the opportunity to successfully undergo this treatment.

In recent years, several groups of investigators have developed non-myeloablative reduced-intensity conditioning (RIC) regimen, which lead to engraftment of donor lymphoid and hematopoietic stem cells without the extra-hematopoietic toxicities of traditional myeloablative transplantations while conserving the GVL or GVT effect after transplantation. This reduced toxicity may make these RIC regimens especially suitable for patients with high-risk of TRM, in particular recipients of second or third transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NB who have failed a prior auto-SCT will be eligible for the present study. Patients should have no severe comorbid organ dysfunction (NCI grade > 2 organ toxicity) at enrollment.

Exclusion Criteria:

* Patients with severe comorbid organ dysfunction (NCI grade > 2 organ toxicity) prior to RIST will be off the present study.
* Patients with progressed tumor prior to RIST will be off the present study.
* Patients whose parents do not want to undergo RIST will be off the present study.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
tumor response, overall survival, event-free survival | from 1 year after reduced-intensity allogeneic hematopoietic stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea